CLINICAL TRIAL: NCT07138131
Title: Impact of Omega 3 in Treatment of Inappropriate Sinus Tachycardia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Yousra Mohsen kamal Ali El -Tabakh, Assistant Lecturer of Pediatrics and Neonatology, Faculty of Medicine, Benha University, Egypt., Benha University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MD 11-4-2023
Record Dates: First submitted 2025-08-16; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Omega 3; Treatment; Inappropriate Sinus Tachycardia
MeSH Terms: interventions — Docosahexaenoic Acids

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Patients received omega-3 supplementation for 3 months.
  Interventions: Drug: Omega 3
- Group B (Active Comparator): Patients received standard follow-up without treatment.
  Interventions: Other: Standard follow-up

INTERVENTIONS:
Drug: Omega 3 — Patients received omega-3 supplementation for 3 months.
  Arms: Group A
Other: Standard follow-up — Patients received standard follow-up without treatment.
  Arms: Group B

SUMMARY:
This study aimed to evaluate the effect of omega-3 supplementation on heart rate (HR) control and heart rate variability (HRV) in children with inappropriate sinus tachycardia (IST).

DETAILED DESCRIPTION:
Inappropriate sinus tachycardia (IST) is a is a common disease of the autonomic nervous system in children in which tachyarrhythmia characterized by a persistent increase in resting sinus rate or disproportionate elevation of heart rate (HR) with minimal physiological effort accompanied by wide ranging symptoms including palpitations, fatigue, presyncope, and exercise intolerance it could cause lead to total disability in severe cases .it also takes a chronic course with Significant adverse effects on quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Age from 12 to 16 years.
* Both sexes.
* Patients diagnosed with inappropriate sinus tachycardia (IST).
* Patients with resting heart rate (HR) ≥100 bpm (sitting) and/or 24-hour average HR ≥90.

Exclusion Criteria:

* Structural heart disease.
* Patients receiving antiarrhythmic medication.
* Patients with a prior history of arrhythmias such as paroxysmal supraventricular tachycardia (PSVT) or sick sinus syndrome, or orthostatic hypotension.
* Secondary conditions such as anemia, infection, or hyperthyroidism.

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Heart rate | 24 hours post-treatment
  Heart rate was recorded at baseline and post-treatment.

SECONDARY OUTCOMES:
Heart rate variability (HRV) | 24 hours post-treatment
  Heart rate variability (HRV) was recorded at baseline and post-treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Benha University, Banhā, Al-Qalyubia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.